CLINICAL TRIAL: NCT01067417
Title: Evaluation of the Efficacy of Hydroxychloroquine in Decreasing Immune Activation in Asymptomatic HIV-infected Patients
Acronym: HCQ-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Collaborators: Wellcome Trust (Other)
Responsible Party: Dr Nick Paton Chief Investigator nip@ctu.mrc.ac.uk, Medical Research Council Clinical Trials Unit
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCQ-01; 2007-005057-36 (EudraCT Number)
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-02

CONDITIONS: HIV Infections
Keywords: Hydroxychloroquine; Chloroquine; HIV Infection; Acquired Immunodeficiency Syndrome; Immune Activation; inflammation; treatment naive; disease progression
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Inflammation; Disease Progression | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxychloroquine (Active Comparator)
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Taken orally 2x200mg capsules once daily for 48 weeks
  Arms: Hydroxychloroquine
Drug: Placebo — Taken orally 2x200mg capsules once daily for 48 weeks
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to find out if taking hydroxychloroquine will decrease immune activation (stimulation of the body's defence system) in people with early HIV infection. Hydroxychloroquine is a medicine that has been used successfully for many years to treat autoimmune diseases (diseases in which the immune system causes damage to the body), e.g. lupus and rheumatoid arthritis. It is generally safe in long-term use and easily accessible.

The immune system is stimulated in response to infections including HIV, so treatments that decrease immune activation may have long-term clinical benefits i.e. delay onset of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV infection on ELISA and confirmatory test.
2. Age 18 to 65 years.
3. Naïve to antiretroviral therapy or off ART for at least 12 months prior to study entry.
4. CD4 T-cell count greater than 400 cells/µL on screening blood test and on one other test performed within the 6 months prior to screening.
5. Plasma HIV RNA viral load greater than 1000 copies/ml on screening blood test
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. History of psoriasis, porphyria cutanea tarda, epilepsy, myasthenia gravis, myopathy of any cause, cardiac arrhythmias, glucose 6-phosphate dehydrogenase (G6PD) deficiency.
2. Insulin-dependent or non-insulin-dependent diabetes mellitus.
3. Chronic liver disease of any cause or alcoholism.
4. Primary HIV infection within 12 months prior to screening, either confirmed (previous negative HIV antibody test within 12 months), or suspected (symptoms strongly suggestive of HIV seroconversion illness within the previous 12 months and patient not known to be HIV antibody positive prior to the illness).
5. Pneumonia, meningitis, septicaemia or any other serious infection in the 2 months prior to screening.
6. Any acute infection with fever and systemic symptoms within the last 24 hours.
7. Any vaccinations in the 2 months prior to screening.
8. Active malignancy (patients are eligible if treatment for the malignancy was completed more than 2 years prior to screening and there has been no subsequent clinical evidence of active disease) or any active immune-mediated or inflammatory disease.
9. Any known suicide attempts (at any time in the past) or current or past history of depression requiring treatment within the 2 years prior to screening. Patients who have not had depression in the previous 2 years but who have had depression in the past may be included if, in the opinion of the physician, the nature of the past episode of depression and the patient's current psychological state indicate that the risk of recurrence of depression during the trial is likely to be low. Patients who have received anti-depressant medication for reasons other than symptomatic depression can be included in the trial.
10. A woman who is currently pregnant or breastfeeding.
11. A woman of child-bearing potential who is planning to become pregnant during the course of the study, or is unwilling to take adequate contraception (including barrier contraception) throughout the course of the study.
12. Use of systemic corticosteroids or other immunomodulatory drugs within the 12 months prior to screening.
13. Current use of medication with known serious hepatotoxic effects or known interaction with hydroxychloroquine.
14. Evidence of cardiac conduction defects or cardiac arrhythmia on screening ECG.
15. Retinopathy or visual field changes detected on screening eye examination.
16. Hepatitis B surface antigen (HBsAg) positive or Hepatitis C PCR positive (patients who are Hepatitis C antibody positive are allowed to participate provided that PCR is negative).
17. Any of the following laboratory abnormalities on screening blood test:

    * Haemoglobin less than 10.5g/dl,
    * Absolute neutrophil count less than 1.0x109/L
    * Platelet count less than 100 X 109/L
    * ALT or AST, or alkaline phosphatase above 2.5 x upper limit of normal (ULN)
    * Serum creatinine greater than 1.5xULN
    * Estimated creatinine clearance (Cockcroft-Gault equation*) below 60ml/min
18. Inability to attend or comply with treatment or follow-up scheduling.
19. Current participation in any other clinical intervention trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-06; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Change in CD8 T-cell activation at week 48 compared to baseline (as shown by a percentage of the cells expressing CD38+ and HLA-DR+). | week 48